CLINICAL TRIAL: NCT02492737
Title: A Phase I, Multicenter, Open-Label, Dose-Escalation and Expansion, Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity Study of Orally Administered AG-881 in Patients With Advanced Hematologic Malignancies With an IDH1 and/or IDH2 Mutation
Brief Title: Study of Orally Administered AG-881 in Patients With Advanced Hematologic Malignancies With an IDH1 and/or IDH2 Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG881-C-001
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome; Hematologic Malignancies
Keywords: acute myeloid leukemia; AML; myelodysplastic syndrome; MDS; dual mutation; MPN; AITL; hematologic malignancies; IDH1; IDH2; AG-881
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AG881 (Experimental): AG-881 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle. Patients may continue treatment with AG-881 until disease progression, development of other unacceptable toxicity or Investigator discretion
  Interventions: Drug: AG881

INTERVENTIONS:
Drug: AG881 — AG-881 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle. Patients may continue treatment with AG-881 until disease progression or development of other unacceptable toxicity

SUMMARY:
The purpose of this Phase I, multicenter study is to evaluate the safety, pharmacokinetics, pharmacodynamics and clinical activity of AG-881 in advanced hematologic malignancies that harbor an IDH1 and/or IDH2 mutation

DETAILED DESCRIPTION:
The first portion of the study is a dose escalation phase where cohorts of patients will receive ascending oral doses of AG-881 to determine maximum tolerated dose (MTD) and/or the recommended Phase II dose. The second portion of the study is a dose expansion phase where patients will receive AG-881 to further evaluate the safety, tolerability, and clinical activity of the recommended Phase II dose. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs or the patient is removed at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

Patients must be ≥18 years of age

Patients must have documented IDH1 and/or IDH2 gene-mutated disease

Patients must have an advanced hematologic malignancy with an IDH1 and/or IDH2 mutation

Patient must be able to understand and willing to sign an informed consent

Patients must have ECOG PS of 0 to 2

Patients must have adequate hepatic function as evidenced by serum total bilirubin ≤1.5 upper limit of normal (ULN), unless considered due to Gilbert's disease or leukemic involvement

Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤3.0 × ULN, unless considered due to involvement by the neoplasm under consideration for treatment

Patients must have adequate renal function as evidenced by a serum creatinine ≤2.0 × ULN or Creatinine clearance 40 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation

Patients must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer

Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of therapy. Patients with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated at all) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

Exclusion Criteria:

Patients who have undergone HSCT within 60 days

Patients who received systemic anticancer therapy or radiotherapy <14 days prior to their first day of study drug administration

Patients who received an investigational agent <14 days prior

Patients who are pregnant or breast feeding

Patients with an active severe infection who require anti-infective therapy or with an unexplained fever >38.5°C during Screening visits or on their first day of study drug administration (at the discretion of the Investigator, patients with tumor fever may be enrolled)

Patients with New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within approximately 28 days of C1D1

Patients with a history of myocardial infarction within the last 6 months

Patients with known unstable or uncontrolled angina pectoris

Patients with a known history of severe and/or uncontrolled ventricular arrhythmias

Patients with QTc interval ≥450 msec or with other factors that increase the risk of QT prolongation or arrhythmic events

Patients taking medications that are known to prolong the QT interval

Patients with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C

Patients with clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid is only required if there is a clinical suspicion of CNS involvement by leukemia during Screening

Patients with immediately life-threatening, severe complications of hematologic malignancies such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability; incidence of adverse events | Up to 26 weeks, on average
Maximum Tolerated Dose and/or the recommended Phase II dose of AG-881 in patients with advanced hematologic malignancies | Up to 26 weeks, on average

SECONDARY OUTCOMES:
Pharmacokinetics of AG-881 in patients with advanced hematologic malignancies | Up to 26 weeks, on average
Pharmacodynamic levels of AG-881 | Up to 26 weeks, on average
Pharmacodynamic levels of 2-HG | Up to 26 weeks, on average
Clinical Activity according to the 2003 revised IWG criteria for AML, the 2006 modified IWG criteria for MDS, disease-specific response criteria for other hematologic malignancies | Up to 26 weeks, on average

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Aurora, Colorado
  - Chicago, Illinois
  - Boston, Massachusetts
  - New York, New York
  - Houston, Texas
- Villejuif, France

REFERENCES:
- [Derived] DiNardo CD, De Botton S, Pollyea DA, Stone RM, Altman JK, Fathi AT, Limsakun T, Liang M, Choe S, Hossain M, Tron AE, Meng Q, Kapsalis SM, Pandya SS, Stein EM. Safety, efficacy, and PK/PD of vorasidenib in previously treated patients with mIDH1/2 hematologic malignancies: A phase 1 study. Am J Hematol. 2023 Sep;98(9):E233-E236. doi: 10.1002/ajh.27005. Epub 2023 Jun 24. No abstract available. PMID 37354069